CLINICAL TRIAL: NCT00739037
Title: A Randomized, Single Dose, Placebo-Controlled, 2 Period Crossover Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PAZ 417 in Cerebrospinal Fluid, When Administered Orally to Subjects With Alzheimer's Disease
Brief Title: Study Evaluating PAZ-417 in Cerebrospinal Fluid in Subjects With Alzheimer's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 3186A1-1103
Record Dates: First submitted 2008-08-15; First posted 2008-08-21 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Experimental)
  Interventions: Drug: PAZ-417

INTERVENTIONS:
Drug: Placebo
  Arms: A
Drug: PAZ-417
  Arms: B

SUMMARY:
The primary purpose of this study is to assess biomarker known as amyloid beta peptide 40 (Ab40) in Cerebrospinal Fluid (CSF), following a single oral dose of PAZ-417 in subjects with Alzheimer Disease (AD). This study will also consider another biomarker amyloid beta peptide 42 (Ab42) in Cerebrospinal Fluid in subjects with Alzheimer Disease and assess the safety, tolerability and pharmacokinetic profile of PAZ-417 in both plasma and Cerebrospinal Fluid in these subjects.

ELIGIBILITY:
Inclusion:

1. Men or women of non-childbearing potential, 55 years of age or older with a probable diagnosis of Alzheimer's Disease (AD), according to the National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria. Subjects will have AD that is mild to moderate in severity, as qualified by a score of 12 to 26 on the Mini-Mental State Examination (MMSE). Woman of non-childbearing potential must be either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal at least 1 year and must have a negative serum pregnancy test result within 48 hours before administration of test article. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue it for 12 weeks after test article administration.
2. Body mass index in the range of 18 to 32 kg/m2 and body weight greater than or equal to 50 kg.
3. Subjects must be generally healthy, with the exception of AD but may be enrolled with a stable, chronic illness, if it is well controlled and does not interfere with the primary objective of the study. Subjects may be included with clinically important deviations from normal limits in medical history, physical examination findings, vital sign measurements, findings on 12 lead electrocardiogram (ECG), or chronic laboratory test results that are associated with stable, well controlled chronic illness.

Exclusion:

1. Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article.
2. Any significant unstable or uncontrolled cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
3. History of vascular disorders (peripheral, coronary, venous), chronic inflammatory disorders (eg, rheumatoid arthritis), hematologic disorders, or bleeding disorders (eg, hemophilia, idiopathic thrombocytopenic purpura, VonWillebrand disease).
4. History of thrombotic events.
5. Presence or history of symptomatic vertigo, significant cardiac valvular disease, congestive heart failure, angina pectoris, significant cardiac arrhythmia, or seizures.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
This study is the measurement of a biomarker known as amyloid beta peptide 40 (Ab40) in Cerebrospinal Fluid (CSF), following a single oral dose of PAZ-417 in subjects with Alzheimer Disease (AD). | 6 days

SECONDARY OUTCOMES:
To measure both amyloid beta peptide 42 (Ab42) and PAZ-417 in both plasma and CSF and assess safety using the results of physical examinations, vital sign measurements, ECGs, cardiac telemetry, standard laboratory tests and collection of AES. | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- California Clinical Trials, Glendale, California, United States